CLINICAL TRIAL: NCT01787136
Title: Dextromethorphan Added on Methylphenidate in the Treatment of the Patients With ADHD
Brief Title: Dextromethorphan Added on for the Patients With ADHD
Acronym: DAOFTPWA
Status: No longer available | Type: Expanded Access
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Chin-Bin Yeh, MD, PhD, Attending Physician, Tri-Service General Hospital
Other Study IDs: TSGH-C97-87
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2022-04-29 (Actual); Status verified 2021-03

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Dextromethorphan

INTERVENTIONS:
Drug: Dextromethorphan — added on therapy
  Other Names: regrow

SUMMARY:
Dextromethorphan added on methylphenidate for the patients with attention deficit hyperactivity disorder

DETAILED DESCRIPTION:
Objectives: Methylphenidate (MPH) is highly effective in controlling the symptoms of attention-deficit/hyperactivity disorder (ADHD), but some children with ADHD either do not respond to, or do not tolerate, treatment. Dextromethorphan (DM) is a neuroprotective agent which has been used in the treatment of neuropsychiatric disorders. This clinical trial had examined the effect of DM on the use of MPH in the children with ADHD.

Methods: This randomized double-blind clinical trial had evaluated 44 male outpatients, aged between 6 and 12 years, with a diagnosis of ADHD. The study subjects were randomly assigned into one of the two groups: receiving MPH alone (15-60 mg per day) or MPH plus DM (30-60 mg per day) for 8 weeks. Assessments, comprising the Chinese version of the Child Behavior Checklist (CBCL-C) scale and the Swanson, Nolan and Pelham Questionnaire (SNAP)-IV rating tests conducted by parents and the serum cytokines measured by microarray and enzyme-linked immunosorband assay (ELISA), were compared between groups at baseline and at 8 weeks after the medication was started.

Results: There were a significant decrease at the mean scores of both CBCL-C and SNAP-IV scales after 8 weeks of treatment, but no significant differences between MPH and MPH+DM groups. Compared with the MPH-only group, the mean scores of some psychometric parameters reported on the CBCL-C and SNAP-IV scales regarding time effects as well as the attention problems on the CBCL-C scale regarding group effect were significantly higher in the DM+MPH group. Although there were no significant differences in the levels of various serum cytokines between groups, the subjects in the DM-MPH group had relatively fewer and lower levels of adverse effects. Significant interactions were found between the withdrawn/depression item reported on the CBCL-C scale and tumor necrosis factor α (ခTNF-α) (p = 0.027), as well as between thought problems item on the CBCL-C and TNF-α (p = 0.028) in subjects who had received DM+MPH treatment.

Conclusion: Following the trial, DM+MPH was not superior to MPH alone for the treatment of children with ADHD, yet DM may potentially have negative effects on ADHD symptoms when combined with MPH.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 6 to 25 who have ADHD symptoms will be recruited. They will be screened for the ADHD symptoms with SNAP 4th version. They then will be referred to a psychiatrist to make a final diagnosis of ADHD by the American Diagnostic Statistical Manual 4th version (DSM-IV).

Exclusion Criteria:

* Patients not willing to participate in the study after detailed explanation.
* Patients who could not follow the investigator's instructions
* Patients who have severe neurological or mental illness like epileptic disorder, history of stroke, schizophrenia, bipolar disorder, mental retardation or uncontrolled suicide risk.
* Patients who have severe medical illness or surgical conditions like uncontrolled abnormal thyroid function, history of heart attack, uncontrolled hypertension.
* Patients who are taking antidepressants, psychotropic medicines within two months prior to the evaluation for entering our study.
* Patients who are allergic to methylphenidate or dextromethorphan.
* Patients with autoimmune disorders
* Patients with asthma or severe infection disorder currently or in the previous two months to avoid the influence of the level of cytokines.

Ages: 6 Years to 25 Years | Sex: All
Age Groups: Child, Adult

REFERENCES:
- [Derived] Chuang WC, Yeh CB, Wang SC, Pan PY, Shyu JF, Liu YP, Gau SS, Lu RB. Potential Negative Effects of Dextromethorphan as an Add-On Therapy to Methylphenidate in Children With ADHD. Front Psychiatry. 2019 Jun 26;10:437. doi: 10.3389/fpsyt.2019.00437. eCollection 2019. PMID 31333511